CLINICAL TRIAL: NCT07154108
Title: A Phase I, Open-label, Two-cohort Study of Recombinant Human Endostatin Adenovirus in Combination With Immune Checkpoint Inhibitors in Patients With Recurrent or Metastatic Head and Neck Cancer or Esophageal Squamous Cell Carcinoma
Brief Title: Endostatin Adenovirus With Checkpoint Inhibitor in Advanced Head and Neck or Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AdEndo-PD1-P1
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Cancer; Head and Neck Cancer (H&Amp;Amp;Amp;N)
Keywords: Esophageal cancer; Esophageal squamous cell carcinoma; Head and neck cancer; Endostatin Adenovirus; safety; Clinical efficacy
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: * Cohort A (Head and Neck Cancer): Patients with recurrent or metastatic head and neck cancer; single-arm, open-label; N ≈ 20
  * Cohort B (Esophageal Squamous Cell Carcinoma): Patients with superficial lymph node metastasis of ESCC; single-arm, open-label; N ≈ 20
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostatin Adenovirus+PD-1 inhibitor (Experimental): Recombinant Human Endostatin Adenovirus: Administered via intratumoral injection twice every 3 weeks for a total of eight doses, or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first. Immune checkpoint inhibitor: Administered via intravenous infusion once every 3 weeks.
  (This study includes two parallel cohorts: Cohort A (recurrent/metastatic head and neck cancer) and Cohort B (esophageal squamous cell carcinoma). Both cohorts will receive the same intervention.)
  Interventions: Biological: recombinant human endostatin adenovirus; Drug: PD-1 Inhibitor

INTERVENTIONS:
Biological: recombinant human endostatin adenovirus — Recombinant Human Endostatin Adenovirus: Administered via intratumoral injection twice every 3 weeks for a total of eight doses, or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first.
Drug: PD-1 Inhibitor — PD-1 inhibitor: Administered via intravenous infusion once every 3 weeks.

SUMMARY:
This is a Phase I, open-label, dual-cohort clinical trial designed to evaluate the safety, tolerability, and preliminary efficacy of intratumoral injection of recombinant human endostatin adenovirus in combination with a PD-1 inhibitor in patients with recurrent or metastatic head and neck cancer, or in patients with esophageal squamous cell carcinoma (ESCC) with superficial lymph node metastasis.

DETAILED DESCRIPTION:
Cohort A will enroll patients with recurrent or metastatic head and neck cancer. Cohort B will enroll patients with ESCC with superficial lymph node metastasis. Both cohorts will receive intratumoral injection of recombinant human endostatin adenovirus combined with intravenous an immune checkpoint inhibitor.

The primary objectives are to assess the safety profile, incidence of dose-limiting toxicities (DLTs), and treatment-related adverse events (TRAEs) of the combination therapy. The secondary objectives include evaluation of objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS). Each cohort plans to enroll approximately 20 patients, with a total of 40 participants.

ELIGIBILITY:
* Cohort A (Head and Neck Cancer)
* Cohort B (Esophageal Squamous Cell Carcinoma)

Inclusion Criteria:

1. Age ≥18 years

   * Cohort A (Head and Neck Cancer): ≤70 years
   * Cohort B (Esophageal Squamous Cell Carcinoma): ≤75 years
2. Histologically or cytologically confirmed recurrent or metastatic:

   * Cohort A: Head and Neck Cancer
   * Cohort B: ESCC, AJCC 9th edition stage IV
3. Prior treatment:

   * Cohort A: ≥1 prior platinum-based chemotherapy regimen or platinum-refractory/intolerant
   * Cohort B: Prior immune checkpoint inhibitor (ICI) therapy with documented acquired resistance after prior PR or SD
4. At least one lesion accessible for intratumoral injection

   * Cohort A: measurable lesion ≥2 cm by RECIST 1.1
   * Cohort B: superficial metastatic lymph nodes (cervical or supraclavicular)
5. ECOG performance status

   * Cohort A: 0-2
   * Cohort B: 0-1
6. Adequate organ function
7. Life expectancy ≥12 weeks (Cohort A)
8. No anti-tumor therapy (chemotherapy, radiotherapy, biotherapy, antiviral) within 4 weeks prior to enrollment (Cohort A)
9. Availability of fresh tumor tissue specimen or pathological slides from the injection target lesion (Cohort B)
10. Male/female patients of childbearing potential must use effective contraception during study and for at least 6 months after treatment
11. Voluntary participation with signed informed consent

Exclusion Criteria:

1. Known allergy or hypersensitivity to study drugs
2. Lesions unsuitable for injection due to proximity to major blood vessels, nerves, or hollow organs, or with extensive necrosis
3. Deeply located lesions with high procedural difficulty (Cohort B)
4. Concurrent radiotherapy to target lesion(s) (Cohort A)
5. Prior anti-angiogenic therapy (Cohort A)
6. Immunosuppressive therapy or systemic corticosteroids >10 mg/day prednisone (or equivalent) within 2 weeks prior to enrollment
7. Active autoimmune disease or history of autoimmune disease
8. Congenital or acquired immunodeficiency
9. Severe coagulopathy, bleeding tendency, or high-risk lesions (Cohort B)
10. Poor nutritional status (Cohort B)
11. Interstitial lung disease with symptoms or radiographic evidence (Cohort B)
12. Severe uncontrolled systemic disease or recent myocardial infarction (<3 months)
13. Acute infection
14. Pregnancy or breastfeeding
15. Other malignancy besides ESCC (Cohort B)
16. Patients unlikely to comply with follow-up or participation requirements
17. Any condition deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse effects (TRAEs) | Through study completion, an average of 1.5 year
  This study will collected any adverse medical events that occurred during the study drug treatment, and the treatment related adverse events as assessed by CTCAE v5.0.
Incidence of Dose-Limiting Toxicities (DLTs) | During the first cycle of treatment （21 days）
  DLTs are defined as treatment-related adverse events occurring during the DLT evaluation period that meet protocol-specified criteria for severity and duration, as assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months
  It is defined as the proportion of patients with complete response (CR) or partial response (PR), as assessed by RECIST 1.1.
Disease Control Rate (DCR) | up to 12 months
  DCR refers to the proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) for a specified minimum duration after treatment, based on RECIST 1.1.
Progression-Free Survival (PFS) | up to 12 months
  Time from the start of treatment to the first documentation of disease progression based on RECIST 1.1.
Overall Survival (OS) | up to 24 months
  Time from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No